CLINICAL TRIAL: NCT04737590
Title: A Randomized Clinical Trial Comparing Curettage With Allogenic Bone Grafting and Curettage With Bioactive Glass Filling in Children With Bone Cysts CYSTS
Brief Title: Bioactive Glass or Allogenic Bone in Pediatric Bone Cysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Bonalive Biomaterials Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2020-12-11; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Bone Cysts
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive glass (Active Comparator): 20 bone cysts (in 20 patients) are filled with bioactive glass
  Interventions: Device: Bioactive glass
- Allogenic bone (Active Comparator): 20 bone cysts (in 20 patients) are filled with allogenic bone
  Interventions: Device: Bioactive glass

INTERVENTIONS:
Device: Bioactive glass — Comparison of bioactive glass to allogenic bone in pediatric bone cysts

SUMMARY:
The Finnish Paediatric Orthopedic Study Group will perform a prospective, randomized, multicenter, clinical trial comparing two bone substitutes (allograft and bioactive glass, BonAlive®) in treating bone cysts in children (18 years or younger). The trial is carried out in five University Hospitals (Turku, Helsinki, Tampere, Oulu, Kuopio) in Finland.

DETAILED DESCRIPTION:
Twenty patients will be randomized into each group. In all University Hospitals the treatment protocol will be same. Randomization will be performed using a sealed envelope technique.

Before surgery all patients will be examined clinically. After conventional radiographs all patients will be examined with magnetic resonance imaging showing cyst's size, anatomy, location and adjacent structures.

If the aneurysmal bone cyst is large or in difficult location, embolization by the radiologist can be used preoperatively.

Surgical technique:

Surgery will be done by experienced paediatric orthopaedic surgeons. Normal orthopaedic exposures will be used. The cyst is opened so that square window is done to the cortex. A sample to the pathologist is collected, also intraoperative frozen section is used to confirm the diagnosis. A mechanical curettage with use of a curette and a high speed burr is used to inspect the whole cavity. The tumour is resected as thoroughly as possible. After curettage 5% phenol is inserted to the cavity and it is neutralized with saline. Cyst volume is evaluated using saline (ml). Then the cyst is filled with morsellized femoral head allograft or bioactive glass (BG-S53P4) according to randomization. The biggest granule size 2-3,15mm is used for femur, tibia, pelvis and humerus. If the cyst volume is below 10ml in these places then smaller granule size (1-2mm) is chosen. If the cyst is in hand region then the granule size is 0,5-0,8mm. At the end of the operation the window's roof is inserted back. All the time X-ray is used to ensure that the whole cyst is treated properly. Osteosynthesis will be performed whenever it is necessary to prevent a pathological fracture.

After surgery the diagnosis will be confirmed histopathologically.

All patients will receive standard anesthesia.

Postoperatively an X-ray will be taken. Radiographic controls after surgery will be held at 1 Mo, 3 Mo, 6Mo, 12Mo and 24Mo. Three months control and two years control will be accompanied with MRI.

If the cyst is found after a pathologic fracture, the fracture is healed first with the cast +/- traction and MRI will be taken before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected aneurysmatic bone cyst in all areas, not spinal.
2. Other large simple bone cyst in load bearing areas
3. Simple or aneurysmal bone cyst and a pathological fracture in non load-bearing areas

Exclusion Criteria:

1. Malignancy
2. Bone marrow disease
3. Other than aneurysmatic or simple bone cyst
4. A secondary aneurysmal bone cyst (ABC associated with another underlying lesion)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | through study completion, average 2 years
  Cyst's recurrence
Recurrence size | through study completion, average 2 years
  The size of cyst recurrence
Operation time | during the surgery
  Time from the cut to the closure
Blood loss | during the surgery
  Operation's blood loss
Complication | during the surgery
  Complications at the operation
Complication | through study completion, average 2 years
  Complications during follow-up
Hospital Stay | immediately after the surgery
  Number of days spent at the hospital
Cyst-healing grade (Enneking's grading system) | through study completion, average 2 years
  Enneking's grading system (scale 1-3, 1=latent, 2=active, 3=aggressive)
Function (Musculoskeletal society tumor score) | through study completion, average 2 years
  Musculoskeletal society tumor score (scale 0-5, 5=best outcome, 0=worst outcome)
Fracture after operation | through study completion, average 2 years
  Fracture after operation at the filled area in radiograph (yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Helenius, Prof, Study Director — University of Helsinki
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku